CLINICAL TRIAL: NCT05832749
Title: Post-market, Prospective, Randomised, Controlled, Masked Clinical Investigation to Compare the Safety and Efficacy of Ophtesis Bio 3% With a Similar 3% Sodium Hyaluronate OVD (Ophthalmic Viscosurgical Device)
Brief Title: Comparison of the Safety and Efficacy of Ophtesis Bio 3% With a Similar 3% Sodium Hyaluronate OVD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gemini Eye Clinic (Industry)
Responsible Party: Principal Investigator, Dr. Pavel Stodulka, Chief eye surgeon, Gemini Eye Clinic
Other Study IDs: OVD PMCF study
Record Dates: First submitted 2023-02-22; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Bilateral Cataract; Unilateral Cataract
Keywords: cataract; eye surgery; ovd; ophtesis bio; sodium hyaluronate
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Product: Ophtesis Bio 3%: Subjects to receive Ophtesis Bio 3% in one eye
  Interventions: Device: Ophtesis Bio 3% ophthalmic viscosurgical device
- Control Product: Healon Endocoat 3%: Subjects to receive Healon Endocoat 3% in one eye
  Interventions: Device: Healon Endocoat 3% ophthalmic viscosurgical device

INTERVENTIONS:
Device: Ophtesis Bio 3% ophthalmic viscosurgical device — Intraocular surgery of the anterior segment, including cataract extraction and intraocular lens (IOL) implantation. The viscoelastic properties of OphtesisBio 3.0% allow lubrication, support and protection of ocular tissues during ophthalmic surgery. Maintains the depth of the anterior chamber during surgery, allows for efficient manipulation with reduced trauma to the corneal endothelium and other surrounding tissues.
  Groups: Study Product: Ophtesis Bio 3%
Device: Healon Endocoat 3% ophthalmic viscosurgical device — Healon@ EndoCoat OVD is an ophthalmic viscoelastic containing 3% sodium hyaluronate indicated for use as a surgical aid in patients undergoing ophthalmic anterior segment procedures including:
  * Cataract surgery with an intraocular lens
  * Cataract surgery without an intraocular lens
  * Secondary intraocular lens implantation
  Healon@ EndoCoat maintains a deep chamber during anterior segment surgery, aids in tissue manipulation during surgery, enhances visualization during the surgical procedure and protects the corneal endothelium and other ocular tissue. The viscoelasticity of the solution maintains the normal position of the vitreous face and prevents formation of a flat chamber during surgery. It may also be used to coat intraocular lenses and insertion instruments prior to intraocular lens implantation.
  Groups: Control Product: Healon Endocoat 3%

SUMMARY:
Prospective, randomized, subject/evaluator-masked post market clinical study at up to 2 sites at Gemini eye clinic in Czech Republic. Randomization will be done by the eye surgeon. The purpose of this post market clinical trial is to compare the safety and efficacy of Ophtesis Bio 3% with a similar 3% sodium hyaluronate OVD in routine cataract surgery.

DETAILED DESCRIPTION:
The purpose of this clinical study is to evaluate the performance of the Ophtesis Bio 3%. The primary endpoint is the rate of intraocular pressure (IOP) spikes of 30 mmHG or greater at the 7-day postoperative visit. The secondary endpoint will be the rate of user acceptance evaluated using the surgeon questionnaire at the surgery day visit. Other key endpoints will include IOP and IOP change from baseline at the 7-day postoperative visit, rate of inflammation measured using Slip Lamp at the 7-day postoperative visit, and rates of serious and/or device-related adverse events. Number of Subjects/eyes: Up to 296 eyes will be enrolled to achieve approximately 148 operated eyes per group.

ELIGIBILITY:
Inclusion Criteria:

* Cataract for which extraction and posterior intraocular lens (IOL) implantation have been planned for one or both eyes
* Clear intraocular media, other than cataract
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Signed informed consent

Exclusion Criteria:

* Pupil abnormalities (non-reactive, fixed pupils, or abnormally shaped pupils)
* Recent ocular trauma or ocular surgery that is not resolved/stable or may affect visual outcomes or increase risk to the subject
* Use of systemic or ocular medications that may affect IOP
* Known steroid responder
* Ocular hypertension of ≥ 20 mmHg, medically-controlled ocular hypertension (regardless of IOP value), or glaucomatous changes in the optic nerve
* Patient is pregnant, plans to become pregnant, is lactating or has another condition associated with the fluctuation of hormones that could lead to refractive changes
* Concurrent participation or participation within 45 days prior to preoperative visit in any other clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cataract for which extraction and posterior intraocular lens (IOL) implantation have been planned for one or both eyes
Sampling Method: Probability Sample
Enrollment: 296 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | 7 days
  Rate of intraocular pressure (IOP) spikes of 30 mmHG or greater
Surgeon questionnaire | first day
  The rate of user acceptance ten questions that can be answered on a scale from 1 to 5, 1 means the worst, 5 the best

SECONDARY OUTCOMES:
Biomicroscopic Slit-Lamp Exam | Pre-operative visit, 7 days
  Rate of inflammation
IOP change | 7 days
  IOP change from Pre-operative visit at the 7-day postoperative visit
IOP change | first day
  IOP change from Pre-operative to up to 1 hour post op
Dilated fundus exam | Pre-operative visit, after only if medically indicated
  Examination to help assess ocular health
Serious and /or Device-Related Adverse Events | first day, 7 days
  Rates of serious and/or device-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Stodulka, MD, Principal Investigator — Gemini Eye Clinic
Locations (3):
- Czechia (3):
  - Gemini Eye Clinic, Průhonice
  - Gemini Eye Clinic, Vyškov
  - Gemini Eye Clinic, Zlín

IPD SHARING:
Plan to Share IPD: No